CLINICAL TRIAL: NCT01381198
Title: Distal Rectus Femoris Transfer as a Part of Multilevel Surgery in Children With Spastic Diplegia - a Randomized Clinical Trial
Brief Title: Distal Rectus Femoris Transfer as a Part of Multilevel Surgery in Children With Spastic Diplegia
Acronym: RectusTrans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Dr. Thomas Dreher, MD, Orthopaedic Department, Universitiy of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RecRan271/2006
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-01

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; distal rectus femoris transfer; stiff knee gait pattern; gait analysis; single event multilevel surgery; randomized trial; crouch gait
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Distal rectus femoris transfer (Active Comparator): Single-event multilevel surgery with a concomitant distal rectus femoris transfer
  Interventions: Procedure: Distal rectus femoris transfer
- No distal rectus femoris transfer (No Intervention): Single-event multilevel surgery without distal rectus femoris transfer

INTERVENTIONS:
Procedure: Distal rectus femoris transfer — Transfer of the distal rectus femoris tendon to the semitendinosus tendon.
  Other Names: rectus tendon transfer; rectus femoris transfer; rectus transposition
  Arms: Distal rectus femoris transfer

SUMMARY:
The purpose of this study is to evaluate the effects of an additional distal rectus femoris transfer carried out as a part of single-event multilevel surgery in children with spastic diplegic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy
* spastic diplegia
* ambulatory
* stiff knee gait

Exclusion Criteria:

* relevant previous surgery at the legs
* Botulinum-toxin-injections 6 months prior surgery

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2007-06; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Range of knee flexion in swing phase | prior intervention (baseline) and 1 year post intervention

SECONDARY OUTCOMES:
Peak knee flexion in swing phase | prior to intervention (basline) and 1 year post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic Department, University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Dreher T, Gotze M, Wolf SI, Hagmann S, Heitzmann D, Gantz S, Braatz F. Distal rectus femoris transfer as part of multilevel surgery in children with spastic diplegia--a randomized clinical trial. Gait Posture. 2012 Jun;36(2):212-8. doi: 10.1016/j.gaitpost.2012.02.017. Epub 2012 Mar 15. PMID 22425637